## Effect of a tele-rehabilitation programme in children with burns: a randomized controlled trial

## May 31 2022

Dear Sir/Madam.

You and your child are cordially invited to participate in a research project led by XXX, a doctoral candidate at the Department of Rehabilitation Sciences at The Hong Kong Polytechnic University. Approved by the PolyU Institutional Review Board (Ref: HSEARS#########), this study aims to explore the effectiveness of tele-rehabilitation for children with burns to improve the accessibility of rehabilitation.

Consulting with parents, researchers will arrange suitable times to provide home rehabilitation services via WeChat and phone calls. This includes education on burn rehabilitation, scar management guidance, fitting of burn rehabilitation aids, and support for daily living and family adjustment. The 8-week program includes approximately one hour of online guidance and feedback weekly, with about 10 minutes daily for rehabilitation follow-up. Additionally, assessments through questionnaires will be conducted before the study, at 4 weeks, and after 8 weeks.

The information you provide as part of this project is research data. Personal data, which is identifiable information, will not include anonymized data. We minimize the use of personal data in the research, accessible only to researchers and their teams for study purposes. Oversight and/or audits may be conducted by authorized members of The Hong Kong Polytechnic University.

All information related to you will be kept confidential and stored in password-protected documents known only to the researchers, to be retained until 2028. PolyU takes reasonable precautions to prevent the loss, misuse, unauthorized access, or damage to your information.

You have the right to withdraw from the study at any time without any form of penalty. Should you have any questions, you can ask the researchers now or later, even after the study has begun.

We sincerely invite you to participate in this study and contribute to the tele-rehabilitation for children with burns.

For inquiries, feel free to call XX#######. If you have any complaints about the conduct of this research, you may contact the secretary of the PolyU Institutional Review Board in writing at institutional.review.board@polyu.edu.hk.

The success of this study relies on your active participation and support. Thank you for your cooperation!

Doctoral Candidate, Department of Rehabilitation Sciences, The Hong Kong Polytechnic University